CLINICAL TRIAL: NCT03026517
Title: Phase I Trial of Phenformin With Patients With Combination BRAF Inhibitor/MEK Inhibitor in Patients With BRAFV600E/K-mutated Melanoma
Brief Title: Clinical Trial of Phenformin in Combination With BRAF Inhibitor + MEK Inhibitor for Patients With BRAF-mutated Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Massachusetts General Hospital (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-318
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Melanoma
Keywords: Phenformin; Dabrafenib; Trametinib; BRAF/MEKi; 15-318
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib; Phenformin

ARMS (1):
- Dabrafenib, Trametinib & Phenformin (Experimental): This is a multi-institution single-arm phase I trial with an expansion cohort at the MTD of Phenformin, in patients with metastatic BRAFV600E/K mutated melanoma. In the dose escalation phase, cohorts of patients will be treated with standard dose Dabrafenib (150 mg PO BID) plus Trametinib (2 mg PO QD) and increasing doses of Phenformin. In the dose-escalation phase of the trial, both patients who have already been treated with a BRAF and/or MEK inhibitor, and treatment-naïve patients will be eligible. The maximally tolerated Phenformin dose was determined to be 100 mg BID. The dose-expansion cohort will enroll up to 10 patients who are treatment- naïve for BRAF inhibitor. In this cohort, patients may be treated with any of the 3 FDA-approved BRAFi/MEKi combinations: dabrafenib/trametinib, vemurafenib/cobimetinib, or encorafenib/binimetinib.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Phenformin

INTERVENTIONS:
Drug: Dabrafenib
Drug: Trametinib
Drug: Phenformin

SUMMARY:
The purpose of this study is to test whether it is safe to give phenformin with the standard drug combination of one of 3 FDA-approved combinations of BRAF inhibitor + MEK inhibitor which are standard treatments for patients with metastatic melanoma whose melanoma has a mutation in a gene called BRAF.

ELIGIBILITY:
Inclusion Criteria:

* AJCC (2009) stage IV melanoma, or stage III melanoma not curable by surgery and which is progressing or in patients whom neo-adjuvant treatment is deemed acceptable. Patients must have at least 1 target lesion measurable by RECIST 1.1 criteria.
* The melanoma must harbor an activating BRAF V600 mutation. Prior therapy with a BRAF and/or MEK inhibitor is allowed in the dose-escalation phase only. However, patients who discontinued previous RAF inhibitor due to intolerance of the drug rather than due to progression will not be eligible.
* Histologic proof of melanoma reviewed and confirmed by the treating institution. The melanoma must have a documented BRAFV600E or BRAFV600K mutation by genotyping or IHC12 performed by a CLIA certified laboratory. At MSK, the Diagnostic Molecular Pathology laboratory has developed and implemented a targeted capture-based next-generation DNA sequencing assay, MSK-IMPACTTM, to profile all protein-coding exons and selected introns from 410 oncogenes and tumor suppressor genes in formalin-fixed paraffin embedded tissues (Cheng, D.T., et al., J Mol Diagn, 2015. 17(3): p. 251-64). MSK-IMPACTTM has been approved by the NY State Department of Health to be run as a clinical assay in the CLIA-compliant Diagnostic Molecular Pathology laboratory. MSK-IMPACTTM is capable of detecting mutations, copy number alterations, and structural variations. BRAF Exon15 was captured by the MSK-IMPACTTM panel and the c.1799T>A (p.V600E) mutation was fully validated as per NYS requirements. Detailed results of the validation of this mutation were included in the validation package submitted to NY State Department of Health.
* At MGH, samples will be tested using a multiplex polymerase chain reaction (PCR) technology called Anchored Multiplex PCR (AMP) for single nucleotide variant (SNV) and insertion/deletion (indel) detection in genomic DNA using next generation sequencing (NGS). Briefly, genomic DNA was isolated from a formalin-fixed paraffin embedded tumor specimen is sheared with the Covaris M220 instrument, followed by end-repair, adenylation, and ligation with an adapter. A sequencing library targeting hotspots and exons in 39 genes (including BRAF, exons 11 and 15) is generated using two hemi-nested PCR reactions. Illumina MiSeq 2 x 147 base paired-end sequencing results are aligned to the hg19 human genome reference using BWA-MEM (Li H and Durbin R. Bioinformatics 2009;25(14):1754-60). MuTect (Cibulskis K, et al. Nat Biotechnol 2013;31(3):213-9) and a laboratory-developed insertion/deletion analysis algorithm are used for SNV and indel variant detection, respectively. This assay has been validated to detect SNV and indel variants at 5% allelic frequency or higher in target regions with sufficient read coverage. This test was developed, and its performance characteristics were determined by the MGH Center for Integrated Diagnostics.
* Patients must be adequately recovered from surgery, radiation therapy, or any surgical complications prior to enrollment.
* Age ≥ 18 years old.
* ECOG performance status of 0-2.
* The ability to swallow pills and otherwise follow the protocol.
* Patients with treated CNS metastases will be eligible if not symptomatic the CNS disease has been stable for a minium of 6 weeks and the patient requires less than or equal to the equivalent of 2 mg/day of dexamethasone.
* Patients must have adequate organ and marrow function as defined below:

  * Absolute Neutrophil Count ≥1.5 K/mcL
  * Platelets ≥100 K/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * Total Bilirubin ≤ 1.2 X institutional upper limit of normal (ULN) or ≤ 3.0 X institutional ULN if the patient has Gilbert's Syndrome
  * AST (SGOT) and ALT (SGPT) ≤ 1.2 X institutional upper limit of normal (ULN)
  * Creatinine ≤ 1.4 mg/dl

Exclusion Criteria:

* Type I or Type II diabetes
* A history of renal failure (unless recovered for at least 6 months), lactic acidosis, recurrent or severe hypoglycemia, or significant chronic obstructive lung disease. Patients will not be excluded for reversible episodes of elevated creatinine due to hypovolemia.
* Acute or chronic liver or renal disease.
* Concurrent use of hypoglycemic agents or any systemic therapy for melanoma. Palliative limited-field radiation therapy will be allowed
* Current use of a prohibited medication.
* Vemurafenib

  * Avoid inducers and inhibitors of CYP3A4
  * Careful with drugs metabolized by CTP1A2 (Clozapam, olanzapine, fluvoxamine, haloperidol, theophylline, caffeine).
* Encorafenib

  * Avoid inducers and inhibitors of CYP3A4
  * Avoid drugs that increase QTc interval
* Dabrafenib

  * Avoid inducers and inhibitors of CYP3A4 or CYP2CA8 (Refer to Appendix C for specific drugs).
* Presence of conditions that will interfere significantly with the absorption of drugs.
* A history of known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Pregnant and/or lactating women
* A prior or concurrent metastatic second malignancy within 3 years, even if it does not require active therapy. For example, patients with concomitant indolent B-cell malignancies will not be eligible. Patients with a prior resected in-situ or stage I malignancy felt to be cured will be eligible.
* Other uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. New York Heart Association class ≥2 will be an exclusion criterion.
* QTc interval > 500 msec unless a bundle branch block is also present.
* Patients with brain metastases unless they meet the criteria of section 6.1.8.
* Patients currently receiving other anti-melanoma treatment. Toxicities attributable to any prior therapy must have resolved to grade 1 or better prior to enrollment. Grade 2 endocrinopathies, except diabetes, that are ongoing from prior immunotherapy will not exclude the patient as long as the patient is on appropriate replacement doses of hormone.
* Patients receiving steroid treatment exceeding replacement dosing
* In the dose expansion phase of the trial, prior treatment with a BRAF inhibitor will be an exclusion criterion. This includes prior adjuvant dabrafenib/trametinib.

Inclusion of Women and Minorities:

* Both men and women, and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  The Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 will be used to determine treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Postow, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Dalton KM, Lochmann TL, Floros KV, Calbert ML, Kurupi R, Stein GT, McClanaghan J, Murchie E, Egan RK, Greninger P, Dozmorov M, Ramamoorthy S, Puchalapalli M, Hu B, Shock L, Koblinski J, Glod J, Boikos SA, Benes CH, Faber AC. Catastrophic ATP loss underlies a metabolic combination therapy tailored for MYCN-amplified neuroblastoma. Proc Natl Acad Sci U S A. 2021 Mar 30;118(13):e2009620118. doi: 10.1073/pnas.2009620118. PMID 33762304
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm